CLINICAL TRIAL: NCT00953420
Title: Phase II Study of Carboplatin and Docetaxel Followed by Epstein-Barr Virus Cytotoxic T Lymphocytes in Patients With Refractory/Relapsed EBV-positive Nasopharyngeal Carcinoma(CADEN)
Brief Title: Carboplatin and Docetaxel Followed by Epstein-Barr Virus Cytotoxic T Lymphocytes
Acronym: CADEN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Chrystal Louis, Assistant Professor Pediatrics-Hem-Onc Cell & Gene, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25145-CADEN; CADEN (Other: Baylor College of Medicine)
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; Carboplatin; Docetaxel; Epstein-Barr Virus; T Lymphocytes; EBV-CTLs
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Epstein-Barr Virus Infections | interventions — Docetaxel; Carboplatin; Dexamethasone; Calcium Dobesilate; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Chemotherapy and Immunotherapy (Experimental): 1. Docetaxel 60 mg/m2 IV on Day 1
  2. Carboplatin with target AUC of 5 (mg/ml x min) on Day 1
  3. Dexamethasone 5 mg/m2/dose (max of 8 mg/dose) po q hs on Day 0, and q am and hs on Day 1
  4. After cycle 1, subsequent cycles of chemotherapy may start once ANC > 1000 and platelets > 100,000 post nadir
  5. Up to an additional 2 cycles of chemotherapy, given per the above schedule, may be given if the EBV-specific cytotoxic T lymphocytes product is not available after the initial 4 cycles
  Interventions: Drug: Docetaxel; Drug: Carboplatin; Drug: Dexamethasone; Biological: EBV-specific cytotoxic T lymphocytes; Biological: G-CSF or Peg-GCSF

INTERVENTIONS:
Drug: Docetaxel — 60 mg/m2 IV on Day 1
  Other Names: Taxotere
Drug: Carboplatin — Target AUC of 5 (mg/ml x min) on Day 1
  Other Names: Paraplatin
Drug: Dexamethasone — 5 mg/m2/dose (max of 8 mg/dose) po q hs on Day 0, and q am and hs on Day 1
  Other Names: Decadron
Biological: EBV-specific cytotoxic T lymphocytes — 1 x 10e8 cells/m2 IV over 1 to 5 min
  Other Names: EBV-specific cytotoxic T lymphocytes 1 x 10e8 cells/m2 IV
Biological: G-CSF or Peg-GCSF — If needed per dose modification guidelines: Peg-GCSF 0.1 mg/kg ≤ 45 kg; 6 mg for > 45 kg subcutaneous on Day 2 or GCSF 5 mcg/kg/day (max of 600 mcg) subcutaneous to start 24 hours after carboplatin administration until ANC > 2500 cells/ul x 2 days after nadir.
  Other Names: Filgrastim or pegylated filgrastim

SUMMARY:
Patients have a type of cancer called nasopharyngeal carcinoma (NPC) that has either come back or not gone away after the best known standard treatments.

Most patients that respond to chemotherapy once their NPC tumors have come back have been treated with a platinum-based medication like cisplatin. However, since many patients are given cisplatin during their initial treatment for NPC, in this study, they will be treated with another platinum-based chemotherapy medicine that has been used in patients with NPC called carboplatin. In this study, carboplatin will be used in combination with another drug called docetaxel. Other studies in patients with advanced head and neck cancer have shown that docetaxel can cause tumors to respond better and allow patients to survive longer when added to the standard treatments for those diseases.

Some patients with NPC show evidence of infection with the virus that causes infectious mononucleosis, known as the Epstein Barr virus (EBV), before or at the time of their cancer diagnosis. EBV is found in the cancer cells of almost all patients with advanced stage disease, suggesting that it may play a role in causing NPC. Previously, patients have been treated with high-risk NPC using EBV-specific cytotoxic T cells. These cells are grown in the laboratory and taught to recognize and attack EBV infected cells. In the past, patients were either given the cells alone or just after they had received a medication to briefly lower their white blood cell count. In both cases, many patients had their tumors shrink and in some cases completely disappear after being treated with these EBV-specific cytotoxic T cells.

Investigators have now decided to look at how patients with NPC and their tumors respond to the treatment combination of chemotherapy and EBV-CTL. Patients are being asked to participate in this study since the NPC tumor is associated with EBV and has either come back or not responded to standard treatment. This combination of chemotherapy and EBV-CTLs is an investigational treatment not approved by the Food and Drug Administration.

The purpose of this study is to see how relapsed or refractory, EBV-associated NPC tumors respond when treated with carboplatin and docetaxel followed by EBV-CTL.

DETAILED DESCRIPTION:
A blood sample will be obtained to start making the CTLs before the patient begins chemotherapy. The patients EBV-specific T cells will be grown while the patient is being treated with chemotherapy and given back to the patient after their chemotherapy is completed.

To prepare the CTLs, 60-70 cc of blood will be taken from the patient. The amount of blood collected depends on their size and weight, no more than 3 cc of blood per kg of body weight will be collected at any one time.

This blood will be used to grow an EBV-infected B-cell line and then a T-cell line. B cells and T cells are types of white blood cells that help fight infections in the body. After growing T cells in the laboratory, these cells will be stimulated with EBV infected B cells. The B cells have been treated with radiation so they cannot grow; however, they can provide the stimulation that will train the T cells to recognize and kill EBV infected cells.

The generation of EBV-CTL requires the use of a special cell line, called lymphoblastoid cell line, which will be made from the blood by infecting cells with EBV. Once the LCLs are made, the T cells will be repeatedly stimulate with the LCLs to make EBV-CTL.

The CTLs will then be tested to make sure they kill the EBV infected cells before they are given back to the patient. If the number of CTLs produced is low, investigators may need to obtain additional blood samples to make these cells.

Because the patients cells are being grown in the laboratory, blood will have to be taken to test for infectious viruses such as hepatitis and HIV and patients will also have to fill in a questionnaire that is given to standard blood donors.

EXPECTED LENGTH OF STUDY The chemotherapy treatment portion is planned as 4 cycles of chemotherapy given every 3 weeks. Up to an additional 2 cycles of chemotherapy may be given if the EBV-CTL product is not available after the initial 4 cycles.

If the patient has been able to complete at least 4 cycles of chemotherapy and the EBV-CTL are ready for infusion,then the cells will be given back to the patient. The infusion of the T cells will last about 1 to 5 minutes after the patient has been pretreated with one dose of Tylenol and Benadryl.

The patient will have another disease re-evaluation 8 weeks after the first EBV-CTL injection. Based upon the patient's response to the first infusion, the patient may receive extra doses of cells if they are available. These would be given every 1.5-3 months. If the patient has additional injections of cells, this will require an additional disease re-evaluation 8 weeks after each infusion.

To learn more about the way the EBV-CTLS are working and how long they last in the body, 10-60 mls of blood will be taken before and after each infusion. Up to 60 ml of blood will also be drawn before each cycle of chemotherapy that occurs at Week 1, Week 4, Week 7, Week 10 before the T cell infusion and then at Weeks 1, 2, 4, 6 and 8 weeks after infusion, and then again at the follow-up visits 5, 8, and 11-12 months after infusion. This blood will be used to look at the immune response to the patient's cancer. If the patient only has one EBV-CTL infusion, up to 108 teaspoons of blood will be drawn to allow for evaluation of his or her response to treatment; however, the total amount of blood collected on this study will depend on the total number of EBV-CTL infusions that the patient has.

The patient and his/her response to therapy will be followed for at least 1 year after treatment on this study ends.

STUDY TREATMENT While the cells are being grown, the patient will be started on chemotherapy in order to shrink the size and/or amount of his/her tumor.

The patient will be treated with a combination of docetaxel and carboplatin chemotherapy. The chemotherapy will be given outpatient over several hours. Docetaxel can cause the body to hold on to extra fluid (fluid retention). This side effect can be prevented in most people if they take a small steroid dose before and after docetaxel is given. Therefore, the night before and on the morning chemotherapy is to start, the patient will take a steroid called dexamethasone by mouth.

Once the patient gets to clinic, he/she will be given a dose of docetaxel and then a dose of carboplatin. Each of these medications will be given into the vein after an IV is placed or into the central line. The patient will then take the last dose of dexamethasone before going to bed that night. The patient will receive chemotherapy treatment once every 21 days as long as the patient's blood counts and laboratory tests have returned to an acceptable level. The patient will have a re-evaluation of his/her disease with imaging scans and laboratory tests after the second round of chemotherapy. If the patient's tumor has not gotten worse and/or has not had severe side effects from the chemotherapy, the patient will be treated with 2 to 4 additional rounds of chemotherapy while we are waiting for the EBV-CTLs to be finished.

The combination of chemotherapy agents used in this study might cause the patient's white blood cells to be low. If they are low for a long period of time or the patient develop a serious infection while they are low, her/she may be given an extra medication called Granulocyte colony-stimulating factor (GCSF). GCSF helps to stimulate the production of white blood cells. However, it is anticipated that most people on the study will not require GCSF.

Once the EBV-CTLs are ready and the patient has recovered from the last round of chemotherapy, the EBV-CTL infusion will be scheduled. The CTL infusion will take place at either Houston Methodist Hospital or Texas Children's Hospital. The CTL infusion takes about 1 to 5 minutes, but patients are typically monitored for up to 4 hours after the infusion to make sure that he/she does not have a reaction to the cells.

END OF TREATMENT AND FOLLOW-UP

The patient will have a number of tests and procedures as part of follow up to treatment. These tests will be used to watch for improvements in tumor size, monitor for side effects from the treatment, evaluate how the T cells are working, and look for any signs that the cancer has come back. The patient's will have a physical exam and standard lab tests, including blood tests, and imaging studies about every 3 months during the first year after treatment.

ELIGIBILITY:
INCLUSION CRITERIA:

* Nasopharyngeal Carcinoma in first or subsequent relapse or with primary refractory disease in whom the EBV-genome or antigens have been demonstrated in tissue biopsy samples
* Age 10 years or older
* Life expectancy of 8 weeks or more
* Karnofsky or Lansky score of 50 or more
* Normal bilirubin level (per institutional standard)
* AST and ALT 1.5 x or less upper limit of normal
* Alk Phos level less than 2.5 x upper limit of normal
* ANC greater than 1500 cells/ul
* Hgb 8.0 or greater
* Platelets 100,000 cells/ul or more
* Creatinine 2 x or less ULN or GFR 50 ml/min/1.73 m2 or more
* Women of child-bearing potential must take/use effective birth control while participating in the study.

EXCLUSION CRITERIA:

* Due to the unknown effects of this therapy on a fetus, pregnant women will be excluded from this research.
* Prior allergic reaction to the study drugs used in this protocol or other drugs formulated with polysorbate 80.
* Known HIV positive subjects since treatment may be significantly immunosuppressive
* Women who are breast-feeding
* Severe intercurrent infection
* Patients, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2014-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is to evaluate the overall response rate for patients with advanced-stage, relapsed/refractory, EBV positive nasopharyngeal carcinoma after re-induction chemotherapy and immunotherapy. | 3 months
  The overall response rate for patients with advanced-stage, relapsed/refractory, EBV positive nasopharyngeal carcinoma after re-induction chemotherapy (treatment with docetaxel and carboplatin) followed by immunotherapy with EBV-specific Cytotoxic T lymphocytes will be measured. Response rates will be estimated as the percent of patients whose best response is a CR or PR, and a 95% confidence interval will be calculated for the fraction of responses obtained.To measure the overall response rate, disease will be determined by imaging (MRI, CT, and/or PET imaging) 8 weeks after immunotherapy. In addition, per standard of care, disease re-evaluation will continue 3 months during the first year after participation and then as clinically indicated per the patient's primary oncologist.

SECONDARY OUTCOMES:
Response to re-induction chemotherapy | 8 weeks
Evaluation of immune response by measuring EBV-DNA levels | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chrystal U Louis, MD, MPH, Principal Investigator — Texas Children's Hospital; Baylor College of Medicine
Locations (3):
- United States (3):
  - Houston Methodist Hospital, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas